CLINICAL TRIAL: NCT02962076
Title: Cardiac Positron Emission Tomography for Detection of Cardiac Sympathetic Dysinnervation to Guide Ablation of Ventricular Tachycardia
Brief Title: Study of Cardiac PET/CT Imaging to Guide Ablation Treatment of Ventricular Tachycardia
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Investigator departing institution and enrollment not met.
Sponsor: Khaled Awad, MD (Other)
Collaborators: Biosense Webster, Inc. (Industry); Washington University School of Medicine (Other)
Responsible Party: Sponsor-Investigator, Khaled Awad, MD, MD, Mercy Research
Organization: Mercy Research (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: F141013002
Record Dates: First submitted 2016-11-09; First posted 2016-11-11 (Estimated); Results first posted 2024-12-24 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-11

CONDITIONS: Ventricular Tachycardia
MeSH Terms: conditions — Tachycardia, Ventricular | interventions — 3-alpha-Hydroxysteroid Dehydrogenase (B-Specific)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Arm - PET/CT Imaging With [C-11] MHED (Experimental): Single Arm - positron emission tomography/computed tomography imaging with [C-11] meta-Hydroxyephedrine tracer
  Interventions: Drug: [C-11] Meta-hydroxyephedrine radioactive tracer (MHED)

INTERVENTIONS:
Drug: [C-11] Meta-hydroxyephedrine radioactive tracer (MHED) — this tracer detects the distribution of sympathetic nerve fibers in the left ventricle

SUMMARY:
Imaging is to be performed prior to procedure using positron emission tomography/ computed tomography (PET/CT), after a special dye is injected. The scans are going to be merged with other cardiac scans when doing the ablation procedure to correlate anatomy with physiology.

ELIGIBILITY:
Inclusion Criteria:

* Clinical indication for ventricular tachycardia (VT) ablation (at least one clinical episode of sustained VT) despite antiarrhythmic drug therapy, or if the patient does not wish to be on one
* Ischemic or nonischemic cardiomyopathy
* Sustained monomorphic VT

Exclusion Criteria:

* Right ventricular VT
* Polymorphic VT or ventricular fibrillation (VF) being the sole detected clinical arrhythmia
* Patient is unable to sign informed consent
* Recent myocardial infarction less than 30 days
* Recent ablation for ventricular tachycardia less than 30 days
* Patient is unwilling or unable to cooperate with the study
* Prosthetic mitral or aortic valve
* General contraindications to VT ablation, e.g., major contraindication to anticoagulation therapy, known presence of left ventricular thrombus, reversible causes of VT or VF
* General contraindications to PET imaging, e.g., pregnancy or lactation
* General contraindication to magnetic resonance imaging or to the administration of gadolinium.
* Contraindication to the placement of hemodynamic support devices, i.e. the presence of mechanical valves or lack of adequate vascular access

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2020-09-21 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2024-10-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Mercy Hospital St. Louis, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Arm - PET/CT Imaging With [C-11] MHED: Patients receiving positron emission/computed tomography imaging with [C-11]-meta-hydroxyephedrine (mHED) tracer
Period: Overall Study
Arm/Group | Single Arm - PET/CT Imaging With [C-11] MHED
Started | 11
Completed | 4
Not Completed | 7
Not completed — MHED tracer not available | 5
Not completed — Protocol Violation | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Groups:
- Single Arm - PET/CT Imaging With [C-11] MHED: Patients receiving PET/CT imaging with [C-11] MHED tracer
Arm/Group | Single Arm - PET/CT Imaging With [C-11] MHED
Number analyzed (Participants) | 10
Age, Continuous [Mean (Full Range); unit: years] | 65.3 [40 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Correlation Between PET Data and Electroanatomic Data
Time Frame: 1 week
Population: No outcomes were measured as no patients had complete data.
Arm/Group | Single Arm - PET/CT Imaging With [C-11] MHED
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Single Arm - PET/CT Imaging With [C-11] MHED
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

LIMITATIONS AND CAVEATS:
Overall study data is limited given the study was terminated before reaching the enrollment goal.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol (2023-04-24): https://cdn.clinicaltrials.gov/large-docs/76/NCT02962076/Prot_000.pdf